CLINICAL TRIAL: NCT05862012
Title: A Phase 1, First-in-Human, Multicenter, Open-Label, Dose Escalation and Dose-Expansion Study of Single-Agent ISB 2001 in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of ISB 2001 in Relapsed/Refractory Multiple Myeloma (TRIgnite-1)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ichnos Sciences SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ISB 2001-101
Record Dates: First submitted 2023-05-04; First posted 2023-05-17 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: ISB 2001; Relapsed/refractory multiple myeloma; Open-label; Dose escalation; Dose expansion
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants with R/R MM will be administered ISB 2001 weekly on Days 1, 8, 15, and 22 of each 28-day cycle, with an additional step-up dose in Cycle 1 on Day 4. Treatment cycle duration is 28 days. Participants will receive ISB 2001 until disease progression, unacceptable toxicity occurs, any criterion for stopping the study treatment or participant withdrawal from the study
  Interventions: Drug: ISB 2001
- Part 2: Dose Expansion (Experimental): Dose expansion cohorts will be initiated to further confirm safety and optimal biologically active dose. Participants will receive ISB 2001 until disease progression, unacceptable toxicity occurs, any criterion for stopping the study treatment or participant withdrawal from the study.
  Interventions: Drug: ISB 2001

INTERVENTIONS:
Drug: ISB 2001 — Participants will receive escalating doses of ISB 2001
  Arms: Part 1: Dose Escalation
Drug: ISB 2001 — Participants will receive injection of ISB 2001 as determined in Part 1.
  Arms: Part 2: Dose Expansion

SUMMARY:
This study is a first-in-human, Phase 1, open-label study that will evaluate safety and anti-myeloma activity of ISB 2001 in participants with relapsed/refractory multiple myeloma (R/R MM).

DETAILED DESCRIPTION:
The study will enroll participants with R/R MM that have been treated with immunomodulatory drugs (IMiDs), proteasome inhibitors, and anti-CD38 therapies either in combination or as a single agent and are refractory to, or intolerant of, established therapies known to provide clinical benefit in MM.

The study will be conducted in two parts:

* Part 1: Dose escalation
* Part 2: Dose expansion

Dose escalation will continue until either the maximum tolerated dose (MTD) is defined, the maximum planned dose is reached, or a recommended phase 2 dose (RP2D) is selected. Dose expansion cohorts will be initiated to further confirm safety and optimal biologically active dose. Participants will receive ISB 2001 until disease progression, unacceptable toxicity occurs, any criterion for stopping the study treatment, or participant withdrawal from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with pathologically confirmed MM with measurable M-protein: serum and/or 24 hour urine, serum-free light chains or measurable isolated plasmacytoma
2. Have an Eastern Cooperative Oncology Group (ECOG) performance status score of 2 or less
3. Must have adequate hematologic, hepatic, renal, and cardiac functions

Exclusion Criteria:

1. Active malignant central nervous system involvement
2. Uncontrolled infection requiring systemic antibiotic therapy or other serious infection prior to C1D1
3. History of autoimmune disease requiring systemic immunosuppressive therapy
4. Any concurrent or uncontrolled medical, comorbid, psychiatric or social condition that would limit compliance with study procedures, interfere with the study results, substantially increase the risk of AEs, compromise ability to provide written informed consent or, in the opinion of the Investigator, constitute a hazard for participating in this study.
5. Female subjects who are lactating and breastfeeding or have a positive pregnancy test during the screening period or on Day 1 before first dose of ISB 2001.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Frequency and Severity Of Treatment-Emergent Adverse Events (TEAEs) | Up to 18 months
Number of Dose-Limiting Toxicities (DLT) During the First 28 Days After the First Administration of ISB 2001 (Cycle 1) in Each Cohort (Part 1) | Up to 28 days

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of ISB 2001 in Serum | Up to 28 days
Time to Reach Maximum Concentration (Tmax) of ISB 2001 in Serum | Up to 28 days
Area Under the Concentration Time Curve in Dosing Intervals (AUC0-tau) of ISB 2001 in Serum | Up to 28 days
Area Under the Concentration Time Curve From Zero to Time t (AUC0-t) of ISB 2001 in Serum | Up to 28 days
Percent Incidence of Anti-Drug Antibody (ADA), Neutralizing Antibody (nAb) and Titer of ADA From Baseline Until End-of-Treatment (EOT) | Baseline to 18 months
Overall Response Rate (ORR) Based on International Myeloma Working Group (IMWG) | 18 months
Complete Response Rate (CRR) Based on International Myeloma Working Group (IMWG) | 18 months
Duration of Response (DOR) Based on International Myeloma Working Group (IMWG) | 18 months
Time to Progression (TTP) | 18 months
Time to Next Treatment (TTNT) | 18 months
Time to Response (TTR) | 18 months
Progression Free Survival (PFS) | 18 months
Overall Survival (OS) | 18 months

CONTACTS AND LOCATIONS:
Locations (11):
- United States (5):
  - Standford Cancer Institute, Palo Alto, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Concord Hospital, Concord, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Peter MacCallum Cancer Center, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- HCG Hospital, Bangalore, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carretero-Iglesia L, Hall OJ, Berret J, Pais D, Estoppey C, Chimen M, Monney T, Loyau J, Dreyfus C, Macoin J, Perez C, Menon V, Gruber I, Laurendon A, Caro LN, Gudi GS, Matsuura T, van der Graaf PH, Blein S, Mbow ML, Croasdale-Wood R, Srivastava A, Dyson MR, Matthes T, Kaya Z, Edwards CM, Edwards JR, Maiga S, Pellat-Deceunynck C, Touzeau C, Moreau P, Konto C, Drake A, Zhukovsky EA, Perro M, Pihlgren M. ISB 2001 trispecific T cell engager shows strong tumor cytotoxicity and overcomes immune escape mechanisms of multiple myeloma cells. Nat Cancer. 2024 Oct;5(10):1494-1514. doi: 10.1038/s43018-024-00821-1. Epub 2024 Sep 11. PMID 39261676